CLINICAL TRIAL: NCT03544307
Title: Taekwondo Training Reduces Blood Catecholamine Levels and Arterial Stiffness in Postmenopausal Women With Stage-2 Hypertension
Brief Title: Taekwondo Training and Postmenopausal Women With Stage-2 Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kosin University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Sang-Ho Lee, Principal Investigator, Kosin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TaekwondoMenopause
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Menopause; Hypertension
Keywords: Taekwondo; Menopause; Hypertension; Arterial Stiffness; Blood Catecholamines
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel design with treatment group and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taekwondo Training (Experimental): Taekwondo training was performed 60 minutes/day, 3 days/week for 12-weeks. Exercise intensity was set at 30-40% of heart rate reserve (HRR) and gradually increased to 50-60% over 12 weeks.
  Interventions: Behavioral: Taekwondo training
- Control (No Intervention): Sedentary control asked not to exercise

INTERVENTIONS:
Behavioral: Taekwondo training — Exercise group
  Arms: Taekwondo Training

SUMMARY:
Aging is associated with hormonal imbalances and progressive decreases in arterial health and function. It is crucial to prevent or reduce the negative effects of aging on hormonal balance and the vasculature by implementing appropriate lifestyle interventions, such as exercise training. We examined the effects of a 12-week Taekwondo training program on blood catecholamines, arterial stiffness (pulse wave velocity, PWV), blood pressure (BP), resting heart rate, and muscular strength in postmenopausal women with stage 2 hypertension.

DETAILED DESCRIPTION:
Using a parallel experimental design, participants were randomly assigned to either a Taekwondo exercise training group (n=10) or non-exercising control group (n=10) for 12 weeks.

Participant in the Taekwondo training group trained 3 days/week for 60 minutes per session, and the intensity progressed weekly. Participants in the control group performed no exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with stage-2 hypertension
* Be postmenopausal
* Be between 65 and 85 years old

Exclusion Criteria:

* Known cardiovascular, metabolic or renal diseases
* Physical limitations that prohibit exercise
* Participates in regular exercise

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — gender identity
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Song Park, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Omaha, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taekwondo Training | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taekwondo Training | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (4) | 70 (4) | 70 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 10 | 10 | 20
Blood epinephrine levels [Mean (Standard Deviation); unit: pg/mL] | 43.6 (6.6) | 43.4 (5.1) | 43.5 (5.9)
Blood norepinephrine levels [Mean (Standard Deviation); unit: pg/mL] — norepinephrine
  pg/mL | 268.6 (41.3) | 243.4 (5.1) | 256 (23.2)
Arterial stiffness [Mean (Standard Deviation); unit: m/s] — brachial-to-ankle pulse wave velocity
  m/s | 8.41 (1.0) | 8.27 (0.67) | 8.34 (0.84)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure
  mmHg | 144 (2) | 143 (2) | 144 (2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Diastolic blood pressure
  mmHg | 98 (2) | 99 (2) | 99 (2)
Hand grip strength [Mean (Standard Deviation); unit: kg] — Hand grip strength
  kg | 24 (4) | 25 (4) | 25 (4)
Leg strength [Mean (Standard Deviation); unit: kg] — leg strength
  kg | 39 (6) | 38 (7) | 39 (7)

OUTCOME MEASURES:

1. Primary Outcome: Blood Epinephrine Levels
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
pg/mL | 39.3 (7.1) | 46.2 (4.7)

2. Primary Outcome: Blood Norepinephrine Levels
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
pg/mL | 232.2 (33.7) | 330 (38.2)

3. Secondary Outcome: Arterial Stiffness
Description: Pulse Wave Velocity
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
m/s | 7.67 (1.0) | 8.48 (1.0)

4. Secondary Outcome: Systolic Blood Pressure
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
mmHg | 130 (2) | 142 (2)

5. Secondary Outcome: Hand Grip Strength
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
kilograms (kg) | 27 (3) | 24 (4)

6. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
mmHg | 87 (2) | 97 (2)

7. Secondary Outcome: Leg Strength
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Taekwondo Training | Control
Number analyzed (Participants) | 10 | 10
kilograms (kg) | 41 (7) | 38 (8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Taekwondo Training | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03544307/Prot_SAP_000.pdf